CLINICAL TRIAL: NCT02963350
Title: A Multicenter, Multi-national Open-label Program to Provide BMN 190 to Patients Diagnosed With CLN2 Disease
Status: Approved for marketing | Type: Expanded Access
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 190-502
Record Dates: First submitted 2016-11-09; First posted 2016-11-15 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: CLN2 Disease

INTERVENTIONS:
Drug: BMN190, recombinant human tripeptidyl peptidase-1 (rhTPP1)

SUMMARY:
* To provide access to BMN 190 to patients with CLN2 disease who cannot participate in a clinical trial.
* To collect additional information on the safety and tolerability of BMN 190 administration in patients with CLN2 disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CLN2 disease as confirmed by deficient TPP1 enzyme activity in leukocytes or molecular analysis by identifying 2 known pathogenic mutations. If enzyme analysis is performed by dried blood spot, diagnosis must be confirmed with molecular testing
* Age ≥2 old at the time of informed consent
* Is willing and able to provide written, signed informed consent. Or, in the case of patients under the age of 18 (or other age as defined by regional law or regulation), provide written assent (if required) and have written informed consent, signed by a legally authorized representative, after the nature of the program has been explained, and prior to any program assessments.
* If sexually active, must be willing to use 2 forms of acceptable methods of contraception while participating in the program.
* If female of childbearing potential, must have a negative pregnancy test at Baseline and be willing to have additional pregnancy tests during the program.
* Willing and able to comply with all program procedures.

Exclusion Criteria:

* Another inherited neurologic disease, e.g., other forms of CLN or seizures unrelated to TPPI deficiency/CLN2 disease (patients with febrile seizures may be eligible).
* Has received stem cell, gene therapy, or ERT for CLN2 disease.
* Contraindications for neurosurgery (e.g., congenital heart disease, severe respiratory impairment, or clotting abnormalities).
* Contraindications for MRI scans (e.g., cardiac pacemaker, metal fragment or chip in the eye, aneurysm clip in the brain).
* Episode of generalized motor status epilepticus within 4 weeks before the first infusion.
* Presence of ventricular abnormality (hydrocephalus, malformation).
* Presence of ventricular shunt.
* Has known hypersensitivity to any of the components of BMN 190.
* Currently enrolled or previously enrolled in a clinical study with BMN 190.
* Use of any investigational product or investigational medical device within 30 days prior to Baseline, or requirement for any investigational agent prior to completion of all scheduled program assessments.
* Have travel plans that may interfere with dosing regimen, scheduled program visits and safety monitoring.
* Has a medical condition or extenuating circumstance that, in the opinion of the physician, might compromise the patient's ability to comply with the protocol required testing or procedures or compromise the patient's wellbeing, safety, or clinical interpretability.
* Pregnancy any time during the program; a female patient judged by the physician to be of childbearing potential will be tested for pregnancy.
* A CLN2 combined motor/language score of less than 1 (apply to US only)
* Asymptomatic (symptomatic is defined as having any evidence of neurological involvement attributed to CLN2 disease irrespective of the CLN2 score, including clinical signs and symptoms of disease such as seizures, ataxia, language delay or other developmental delays) (apply to US only)

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cohen Pfeffer, MD, Study Director — Medical Monitor
Locations (5):
- United States (2):
  - Orange, California
  - Columbus, Ohio
- Hamburg, Germany
- Rome, Italy
- London, United Kingdom